CLINICAL TRIAL: NCT07260071
Title: Family Study of Early Hypertension in Children and Young People at Risk of Autosomal Dominant Polycystic Kidney Disease
Brief Title: Hypertension in Children and Young People at Risk of Autosomal Dominant Polycystic Kidney Disease
Acronym: HIYA-PKD
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 347395
Record Dates: First submitted 2025-11-13; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD
Keywords: hypertension; children; young people; autosomal dominant polycystic kidney disease; arterial stiffness; genetic testing; albuminuria; proteinuria
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Hypertension; Albuminuria; Proteinuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADPKD positive: Participants with positive renal MRI and/or genetic test for ADPKD
- ADPKD negative: Participants with negative renal MRI and genetic test for ADPKD

SUMMARY:
The goal of this project is to measure the prevalence of Autosomal Dominant Polycystic Kidney Disease (ADPKD) and hypertension in the general population of children and young people at risk of ADPKD, using magnetic resonance imaging (MRI) for rapid diagnosis alongside genetic testing. The main question it aims to answer is:

What is the prevalence of hypertension in a population sample of adolescents with ADPKD?

Participants will have the following measurements performed:

* Height and weight.
* Blood pressure.
* Non-invasive measurement of arterial stiffness.
* Cardiac and renal MRI.
* Blood sample.
* Genetic testing.

DETAILED DESCRIPTION:
INTRODUCTION Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the commonest genetic cause of chronic kidney disease. Despite being inherited, most people do not get symptoms until adulthood with mean age of chronic renal failure around 53 years. Hence, it was thought that there is no need to screen children and young people (C&YP) at risk of ADPKD until old enough to understand and agree to testing. Linked to this, imaging criteria to diagnose ADPKD mostly cover adult ages.

The validity of this 'adults only' approach is challenged by reports of hypertension in C&YP with ADPKD, affecting up to a quarter by late teens. This is important in deciding whether to change screening policy because early treatment has the potential to reduce risk of cardiovascular events long-term. Death from cardiovascular disease is still a frequent event in ADPKD families, even before reaching end-stage kidney disease. Not only does the renal damage in ADPKD affect BP and cardiovascular health but there is evidence that ADPKD causes generalised endothelial dysfunction. This provides further justification for good BP control and treatment from the earliest stages of ADPKD.

Currently, it is not known whether the estimated prevalence of hypertension in C&YP with ADPKD is overestimated because most evidence comes from specialist Paediatric Nephrology centres, where it would be expected that the more severe cases would be managed. This study will determine whether blood pressure (BP) should be screened in all C&YP at risk, as well as testing the utility of ultrasound and genetic approaches.

This proposed study will be most comprehensive assessment of blood pressure in ADPKD across all age groups. As a result, information gained may revolutionise the approach to the measurement and management of BP in medical practice, particularly in children.

PATIENT AND PUBLIC INVOLVEMENT This study has been set up to specifically consider individuals with ADPKD and so the investigators have designed this study in discussion with The PKD Charity. The investigators will continue to utilise this wealth of patient experience as this study is conducted by keeping the PKD Charity informed of progress, presenting results at patient group meetings and conferences, so that patients are able to see the work that the investigators are doing to improve their understanding of ADPKD. Any publications resulting from this work will be sent to the PKD Charity for inclusion on their website.

A trustee of the PKD charity and patient representative for ADPKD has previously reviewed patient information sheets and consent forms and as a result of helpful comments the investigators have modified the patient information sheet for children.

Lastly these proposals have been previewed as a 'theoretical potential study' on the UK PKD Charity forums: no-one expressed concerns over the study design and over 40 responders expressing immediate interest in participating.

PARTICIPANT SELECTION Source of participants

The study will be advertised on the PKD website, and via social media, leaflets and letters in clinic. This strategy aims to ascertain participants from an unbiased population, to ensure the scientific aims of this study are met which is to determine the true blood pressure levels in C&YP with ADPKD. In addition, using these channels publicises the study without any pressure on families/children to get involved since they have to make the first contact to express interest. Interested participants or their parents/guardians will be able to contact the research team to find out more about the study. Enquiries about study enrolment will be fielded by the Study Co-ordinator, based at King's College London. The study coordinator can ascertain initial eligibility, whilst referring any queries to the Chief Investigator. If the participant appears to be eligible for the study, the relevant Participant Information Sheet (Parent and Adolescent/16+ versions) can be sent out to the participant and their family. The study coordinator will book an appropriate time for the participant and their parent/guardian to attend their most convenient participating site

Number of participating sites involved: 3

Participant numbers: The study aims to recruit 200 C&YP in total. This generates a 95% confidence of detecting a difference between populations with hypertension prevalence of 20% (ADPKD) versus 10% with 80% power. Once they have undertaken the full BP and cardiovascular assessment (anticipated over 1-2 visits), participants will only be seen once and will not be required for further follow up. Results of genetic testing are anticipated to be available after 6-12 months.

STUDY PROCEDURES Screening Procedures

Interested participants or their parents/guardians will be able to contact the research team to find out more about the study. Enquiries about study enrolment will be fielded by the Study Co-ordinator, based at King's College London. The study coordinator can ascertain initial eligibility, whilst referring any queries to the Chief Investigator. If the subject appears to be eligible for the study, the relevant Patient Information Sheet (Parent and Adolescent/16+ versions) can be sent out to the participant and their family. All participants that undergo screening will be logged onto a screening log associated with the study.

Once eligibility is confirmed, and the participant has received the PIS, the study coordinator will contact them to book an appropriate time for the participant and their parent/guardian to attend their most convenient participating site.

Participant recruitment The study will be advertised on the PKD website, and via social media, leaflets and letters in clinic. This strategy aims to ascertain participants from an unbiased population, to ensure the scientific aims of this study are met which is to determine the true blood pressure levels in C&YP with ADPKD. In addition, using these channels publicises the study without any pressure on families/children to get involved since they now have to make the first contact to express interest.

Participants will be offered reimbursement of their reasonable expenses for them and their parent /guardian to attend their chosen participating site.

Participants and their parent/guardian will be sent age appropriate information sheets prior to their first appointment at the hospital and will have at least a week to consider their participation in the study. Written materials will be produced in English. They will be consented by a clinician when they attend for Visit 1 of the study.

Follow up Procedures When the results of the tests are ready, families will be informed of the results with a telephone consultation. If there is no evidence of ADPKD, hypertension or other novel findings, the participant will be discharged. If there is evidence of ADPKD, hypertension or another medical condition, the participant will be followed up in an NHS clinic as per standard of care.

Radiology Assessments MRI will be used to scan the kidneys for evidence of ADPKD and assess the structure and function of the heart. Both regions will be imaged in the same scan session. No contrast will be required.

MRI safety aspects will be handled by the research MRI staff in the study centre. Experienced MRI radiographers will ensure all participants have completed an MRI safety questionnaire prior to their MRI scan as per the Safety Guidelines for Magnetic Resonance Imaging Equipment in Clinical Use, MHRA, February 2021 https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/958486/MRI_guidance_2021-4-03c.pdf.

END OF STUDY DEFINITION

• The date of when all the samples from all patients have been analysed.

ASSESSMENT OF SAFETY

* No particular serious adverse events (SAEs) are expected to occur during this study.
* Where a SAE is related to the study procedures and is an unexpected occurrence (that is, the type of event is not listed in the protocol as an expected occurrence) then it will be reported immediately upon knowledge of the event to R&D and always within 24 hours. A note will be put in the case report form (CRF) and on the participants medical notes.
* If a SAE/AE occurs that does not require immediate reporting, this will be reported in the participant's CRF and reported to GSTT when copied into the Annual Progress Report.
* All serious adverse events that are to be reported to R&D will be signed and dated and completed by the Investigator.
* At other sites, the Principal Investigators at all sites must report all SAEs to the Chief Investigator first where possible. The Chief Investigator is then responsible for reporting events to the regulators/R&D as the sponsor office.

Trial Steering Committee (if applicable) N/A

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 17 years at the time of consent
* Able to tolerate the key study investigations (office blood pressure measurement, ambulatory blood pressure measurement, MRI and blood test)
* Parent with confirmed clinical diagnosis of ADPKD
* Parent (if child <16 years) or both parent and young person (if >=16 years) consents to genetic testing for ADPKD and demonstrates understanding of the implications of this.

Exclusion Criteria:

* 18 years or above at the time of study entry
* Unable to tolerate key study investigations
* Presence of associated co-morbidities which make it difficult to interpret results, including congenital cardiac anomalies and known TSC-PKD1 mutations
* Unwilling to undergo genetic testing for ADPKD

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: General population of children and young people at risk of ADPKD
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with hypertension in general population of children and young people at risk of ADPKD. | Day 1
  Diagnosis of hypertension from clinic manual blood pressure and 24 hours ambulatory blood pressure measurement

SECONDARY OUTCOMES:
Number of participants diagnosed with ADPKD from renal MRI compared to the number from genetic testing. | Day 1
  Prevalence of ADPKD assessed by renal MRI compared to genetic testing
Number of participants with cyst negative but gene positive ADPKD in this age group. | Day 1
  Agreement between MRI and genetic testing for diagnosis of ADPKD.
Number of participants with abnormal albuminuria in the population at risk of ADPKD. | Single time point
  Presence of albuminuria in urine samples collected.
Central blood pressure in young people with ADPKD compared to healthy controls | Day 1
  Comparison between central aortic systolic and diastolic pressure (mmHg) measured by tonometry between participants with ADPKD and healthy controls
Arterial stiffness in young people with ADPKD compared to healthy controls | Day 1
  Comparison in carotid-femoral pulse wave velocity (m/s) between participants with ADPKD and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sinha, PhD, MRCP (UK), MRCPCH, Principal Investigator — King's College London
Locations (1):
- Evelina London Children's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared beyond the study team.

REFERENCES:
- [Background] Ecder T, Schrier RW. Cardiovascular abnormalities in autosomal-dominant polycystic kidney disease. Nat Rev Nephrol. 2009 Apr;5(4):221-8. doi: 10.1038/nrneph.2009.13. PMID 19322187
- [Background] Pei Y, Obaji J, Dupuis A, Paterson AD, Magistroni R, Dicks E, Parfrey P, Cramer B, Coto E, Torra R, San Millan JL, Gibson R, Breuning M, Peters D, Ravine D. Unified criteria for ultrasonographic diagnosis of ADPKD. J Am Soc Nephrol. 2009 Jan;20(1):205-12. doi: 10.1681/ASN.2008050507. Epub 2008 Oct 22. PMID 18945943
- [Background] Torres VE, Harris PC, Pirson Y. Autosomal dominant polycystic kidney disease. Lancet. 2007 Apr 14;369(9569):1287-1301. doi: 10.1016/S0140-6736(07)60601-1. PMID 17434405
- See also: Polycystic Kidney Disease Charity website — https://pkdcharity.org.uk/research/pkd-uk-research/hiya-pkd-study